CLINICAL TRIAL: NCT03521206
Title: Advance Care Planning in Nursing Homes in Flanders, a Cluster Randomized Controlled Trial and Process Evaluation
Brief Title: Advance Care Planning in Nursing Homes in Flanders
Acronym: ACP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: End-of-Life Research Group (Other)
Responsible Party: Principal Investigator, Lieve Van den Block, Professor, End-of-Life Research Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 001
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Advance Care Planning; Elderly Care; Nursing Home
Keywords: Advance directives; Effectiveness; Process evaluation; Care staff

STUDY DESIGN:
Intervention Model Description: Seven of the 14 nursing homes will be randomized to the intervention group. The other seven nursing homes will be randomized to the control group.
Who Masked: Investigator
Masking Description: During the data collection the investigators cannot be blinded, due to the nature of the intervention. However, during data analysis the researchers will be blinded for the unit of randomization of each nursing home, making use of encrypted data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The ACP+ programme aims to improve or establish advance care planning (ACP) in the day-to-day routine of staff working in nursing homes.
  The intervention implementation period has a total duration of 8 months and is divided into:
  * a four-month preparation and training phase. During this phase the ACP reference persons will attend a "two-day training" given by the ACP trainers. Other staff will receive training by the reference persons on conducting ACP conversation or recognizing triggers for an ACP conversation in nursing home residents.
  * A four-month follow-up phase in which ACP conversations are held with residents. Additional training sessions will be organized to give more in-depth knowledge to the ACP reference persons.
  Interventions: Behavioral: ACP+ programme
- Control group (No Intervention): The staff of nursing homes in the control group will receive no additional training next to any standard education or continuous training. After the intervention and follow-up measures are finished, all nursing homes in the control group will be offered a shortened version of the ACP+ training programme as well as all ACP+ training materials.

INTERVENTIONS:
Behavioral: ACP+ programme — Training program for nursing home staff.
  Arms: Intervention group

SUMMARY:
Advance care planning (ACP) is a process that supports adults at any age or stage of health in understanding and sharing their personal values, life goals, and preferences regarding future (medical) care. ACP is of particular relevance for frail older adults, particularly in the nursing home setting where an important proportion of older people die. However, the actual implementation of ACP in nursing home practice seems to be a challenge in many countries worldwide, and people often do not get the opportunity to discuss their preferences in advance. This study evaluates the effectiveness of a theory-based advance care planning training programme (ACP+ programme) for nursing homes in Flanders, Belgium, using a cluster randomised controlled trial (cRCT) design. The ACP+ programme aims to integrate ACP in routine nursing home care by training the nursing home staff and management. Residents and their family will receive in-depth information on ACP and participate in one or several ACP conversations, if they wish so.

Who can participate? Nursing homes that conform to the eligibility criteria: at least 100 beds, situated in Flanders and did not participate in a similar research or implementation project over the last 4 years.

What does the study involve? The researchers will perform a cluster randomized controlled trial (cRCT) to evaluate the effects of an ACP training programme in nursing homes in Flanders (Belgium), accompanied by a process evaluation. Fourteen nursing homes will be randomized to either the intervention group, which will receive the intervention (ACP+ programme), or the control group, in which no additional training regarding ACP (other than that which is part of routine practice) will be provided. The nursing homes in the control group will receive a short training on ACP, as well as all training materials used in the intervention after the last follow-up measurements.

At month 0 the researchers will perform a baseline measurement in the intervention and control groups using structured questionnaires to be filled in by all care staff in the nursing home. At the end of month 8, the same questionnaires will be administered again in all nursing homes (follow-up). The process evaluation will employ structured diaries for ACP trainers, attendance lists for training sessions, audiotaping of a sample of ACP conversations and individual and group interviews with staff and management of the intervention homes.

Hypotheses The primary hypothesis is that the introduction of the ACP+ programme in nursing homes will improve the knowledge and self-efficacy of nursing home care staff regarding advance care planning.

DETAILED DESCRIPTION:
Study hypothesis The primary study hypothesis is that the introduction of the ACP+ programme in nursing homes will improve the knowledge and self-efficacy of nursing home care staff regarding advance care planning (ACP).

Ethics approval The study was approved by the Ethics committee of University Hospital Brussels (Vrije University Brussels, 22/02/2018, ref: 18-003 - B.U.N. 143201834759)

Study design A cluster randomized controlled trial using baseline and follow-up measurement of relevant outcome variables and process evaluation. The trial will be implemented in a sample of 14 nursing homes (see eligibility criteria below) randomised to either intervention or control group.

Trial duration The duration of the entire trial, from the moment the first nursing home is recruited until the end of follow up will be 10 months.

At month 0, immediately after randomization, the baseline assessment is completed in both intervention and control homes. Staff did not know the outcome of the randomisation when filling in the baseline measures (with the exception of the nursing home director).

At month 1, the ACP+ programme will start in nursing homes in the intervention group. This programme consists of two parts, each lasting 4-months (see intervention below for more details), taking up a total of 8 months.

At the end of month 8, follow-up measures will be collected in both groups. The process evaluation will run through the intervention period, starting at month 1 and will be completed at month 9.

Randomisation Paired randomization of nursing homes to the control and intervention groups is performed by an independent and blinded statistician. Criterion is facility status (public vs. private without profit objective vs. private with profit objective).

Sample size calculation Given an expected effect size of d=0.50, the analysis will have power of 80.27% to detect a difference between intervention and control group on the primary outcome (knowledge and self-efficacy of care staff regarding ACP) at follow-up compared to baseline, with a two-sided significance level α=0.025.

Assuming an intra cluster correlation coefficient (ICC) of 0.036, we need to involve at least 161 staff members per study arm. To allow for an initial response rate of 70% and a staff turn-over of 10%, this number is increased to 242 staff members per study arm, 484 members in total. As the average staffing level is 5 FTE for nurses (including 1 FTE head nurse) and 5 FTE for care assistants per 30 beds and the included nursing homes are all required to have over 100 beds, we expect at least 35 care staff members per cluster (nursing home). We will, therefore, need to include 14 nursing homes to achieve the necessary sample of care staff.

Intervention The ACP+ programme is offered in addition to any standard education or continuous training that staff receive in each of the participating nursing homes randomised to the intervention group. Throughout the ACP+ programme, a professional trainer is made available by the research team to train the nursing home staff and to guide implementation of the programme. The ACP+ programme aims to improve or establish advance care planning (ACP) in the day-to-day routine of staff working in nursing homes. At the core of the intervention is the nomination of several representatives for ACP (named ACP reference persons) in each facility who are trained by a specialised ACP trainer made available through the study. During the study period, the specialised trainer will provide training and support to all staff in the nursing homes and specifically support the ACP reference persons in developing their knowledge and skills regarding ACP, implementing the ACP+ programme and training other nursing home staff.

The intervention consists of two parts. The first part focuses on buy-in from management and development of facility-level ACP policy and training staff. A central element is the training of 'ACP reference persons' (who are nurses of the facilities, 3-4 per facility), who will themselves train the other staff in ACP, with the support of the external trainer (train-the-trainer approach). The second part focuses on nursing home staff conducting ACP conversations with residents and family. In addition, the trained staff will be offered more in-depth training sessions (so called 'comeback-seminar' to evaluate the progress they have made so far, and 'specialisation sessions' on handling ACP with residents living with dementia and professional communication) to extend their knowledge and skills, as well as one-on-one coaching.

The intervention implementation period has a total duration of 8 months and is divided into:

* a four-month preparation and training phase. During this phase the ACP reference persons will attend a "two-day training" given by the ACP trainers. Other staff will receive training by the reference persons on conducting ACP conversation or recognizing triggers for an ACP conversation in nursing home residents.
* A four-month follow-up phase in which ACP conversations are held with residents. Additional training sessions will be organized to give more in-depth knowledge to the ACP reference persons.

The staff of nursing homes in the control group will receive no additional training next to any standard education or continuous training. After the intervention and follow-up measures are finished, all nursing homes in the control group will be offered a shortened version of the ACP+ training programme as well as all ACP+ training materials.

Statistical analysis The researchers will conduct regression analyses to test study hypotheses using intention-to-treat (ITT) and per protocol approaches. Multi-level mixed model regression analyses will be used to analyze outcomes, controlling for baseline values and clustering of data within the nursing homes. Within the multi-level mixed model analyses, outcomes will be analyzed with nursing homes as random factor, and group, time point, and their interaction as fixed factors. Differences in mean change between the intervention group and the control group (group by time interaction) will be calculated. The effect sizes (Cohen's d) using the baseline-adjusted mean differences and the variance between nursing home staff and between nursing homes will be estimated to assess effect sizes for the different outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for nursing homes:

  1. the board of directors/the management express explicit motivation to participate in the study and agree to allocate at least a 0,10 FTE per week for at least two ACP Reference Person(s) per 30 to 40 nursing home beds, to carry out the tasks that are part of this project
  2. have at least 100 beds

Inclusion criteria for care staff in the nursing homes:

1. able to speak and understand Dutch.
2. work in a participating nursing home as either (head) nurse, care assistant, psychologist, physiotherapist, occupational therapist, social worker, animator, or reference person dementia/palliative care

Exclusion Criteria:

* Exclusion criteria for nursing homes:

  1. nursing homes have taken/are taking part in another research study that is evaluating palliative care services or communication strategies, currently or in the past 4 years
  2. they have - or are planning to develop during the foreseen duration of the trial - an extensive ACP policy, meaning that (i) all nursing home residents or their family (in principal) regularly receive ACP conversations (two conversations or more each year) or (ii) the nursing home is judged by the researchers as having explicit and detailed ACP guidelines available (corresponding to high-quality ACP procedures and practices)
  3. major organisational changes or physical changes to the facility (e.g. building activities or staff re-organisation) are planned or ongoing during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of and self-efficacy concerning ACP | One questionnaire at baseline (T0), one questionnaire at follow-up (T1, 8 months after T0)
  The knowledge questions concern legal rules and regulations in Belgium around ACP-related issues (for example, the legal status of an advanced directive). The self-efficacy questions survey the respondent's self-efficacy regarding ACP.

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Van den Block, Prof. Dr., Principal Investigator — VUB
Locations (1):
- End of Life Care Research Group, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivodic L, Wendrich-van Dael A, Gilissen J, De Buyser S, Deliens L, Gastmans C, Vander Stichele R, Van den Block L. Effects of a theory-based advance care planning intervention for nursing homes: A cluster randomized controlled trial. Palliat Med. 2022 Jul;36(7):1059-1071. doi: 10.1177/02692163221102000. PMID 35769038
- [Derived] Gilissen J, Wendrich-van Dael A, Gastmans C, Vander Stichele R, Deliens L, Detering K, Van den Block L, Pivodic L. Differences in advance care planning among nursing home care staff. Nurs Ethics. 2021 Nov-Dec;28(7-8):1210-1227. doi: 10.1177/0969733021994187. Epub 2021 May 5. PMID 33947293
- [Derived] Gilissen J, Pivodic L, Wendrich-van Dael A, Cools W, Vander Stichele R, Van den Block L, Deliens L, Gastmans C. Nurses' self-efficacy, rather than their knowledge, is associated with their engagement in advance care planning in nursing homes: A survey study. Palliat Med. 2020 Jul;34(7):917-924. doi: 10.1177/0269216320916158. Epub 2020 May 8. PMID 32383636
- [Derived] Gilissen J, Pivodic L, Wendrich-van Dael A, Gastmans C, Vander Stichele R, Engels Y, Vernooij-Dassen M, Deliens L, Van den Block L. Implementing the theory-based advance care planning ACP+ programme for nursing homes: study protocol for a cluster randomised controlled trial and process evaluation. BMC Palliat Care. 2020 Jan 8;19(1):5. doi: 10.1186/s12904-019-0505-7. PMID 31915000